CLINICAL TRIAL: NCT02713191
Title: Efficacy and Safety of Dexmedetomidine vs. Midazolam Sedation in Patients Undergoing Convex-probe Endobronchial Ultrasound: a Randomized Double Blind Trial
Brief Title: Dexmedetomidine vs. Midazolam Sedation for Endobronchial Ultrasound
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashutosh Nath Aggarwal, Professor of Pulmonary Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Renu1
Record Dates: First submitted 2016-01-20; First posted 2016-03-18 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Conscious Sedation During Procedure; Endobronchial Ultrasound
Keywords: Bronchoscopy; Sedation; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine + fentanyl before, and dexmedetomidine infusion during, procedure
  Interventions: Drug: Dexmedetomidine; Drug: Rescue midazolam; Drug: Fentanyl
- Midazolam (Active Comparator): Midazolam + fentanyl before, and matching saline infusion during, procedure
  Interventions: Drug: Midazolam bolus; Other: Saline placebo; Drug: Rescue midazolam; Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 1µg/Kg in 100 mL saline intravenously over 10-15 minutes immediately prior to procedure, followed by Dexmedetomidine infusion at 0.6 µg/kg/hour as maintenance dose during entire procedure
  Arms: Dexmedetomidine
Drug: Midazolam bolus — Midazolam 2 mg as slow intravenous bolus immediately prior to procedure
  Arms: Midazolam
Other: Saline placebo — 100 mL saline infusion over 10-15 minutes immediately prior to procedure
  Arms: Midazolam
Drug: Rescue midazolam — Rescue boluses of 0.5 mg midazolam, if needed during procedure
Drug: Fentanyl — 1 µg/kg fentanyl as slow intravenous bolus immediately prior to procedure

SUMMARY:
The randomized controlled trial will compare efficacy and safety of dexmedetomidine to midazolam for sedation during endobronchial ultrasound

DETAILED DESCRIPTION:
Benzodiazepines, opioids, and propofol are currently used alone or in combination for achieving sedation during endobronchial ultrasound and other bronchoscopic procedures. However, all these agents carry a risk of respiratory depression. Dexmedetomidine, a highly selective adrenergic alpha-2 agonist, has sedative and analgesic properties but does not cause respiratory depression. This study aims to compare efficacy and safety of dexmedetomidine as a sedative to midazolam in patients with hilar/mediastinal lymphadenopathy undergoing convex-probe endobronchial ultrasonography on day care basis. Patients will be randomized to receive either dexmedetomidine plus fentanyl or midazolam plus fentanyl prior to procedure, followed by dexmedetomidine or saline infusion respectively during the procedure. Ramsay sedation score of two will be targeted, failing which patients in both groups will receive midazolam bolus on as-needed basis. Bronchoscopist will remain blinded to group allocation. Patients will be monitored for sedation, oxygenation and hemodynamic parameters throughout. Need for additional midazolam, sedative efficacy, frequency of adverse respiratory and hemodynamic events, and bronchoscopist and patient satisfaction with the procedure will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* American Society of Anesthesiologists physical status I or II
* Presence of hilar and/or mediastinal lymph nodes on thoracic CT scan

Exclusion Criteria:

* Known allergy to dexmedetomidine or midazolam or fentanyl
* Documented coagulopathy
* Pregnancy
* Hemodynamic instability (hypotension, arrhythmia, recent acute coronary event)
* Neuropsychiatric illness
* History of previous endobronchial ultrasound procedure
* Refusal to provide consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Number of midazolam boluses administered to achieve targeted Ramsay sedation score of two | From start of endobronchial ultrasound procedure until finish of endobronchial ultrasound procedure, assessed up to two hours

SECONDARY OUTCOMES:
Mean difference in depth of sedation during procedure as assessed by Ramsay scale | From start of endobronchial ultrasound procedure until finish of endobronchial ultrasound procedure, assessed up to two hours
Frequency of adverse hemodynamic events - hypotension, hypertension, tachycardia, bradycardia | From start of endobronchial ultrasound procedure until finish of endobronchial ultrasound procedure, assessed up to two hours
Frequency of respiratory events - hypoxia, need for air airway maneuvers to maintain oxygenation | From start of endobronchial ultrasound procedure until finish of endobronchial ultrasound procedure, assessed up to two hours
Mean difference in patient and physician satisfaction related to procedure as assessed by visual analogue scale | Immediately after endobronchial ultrasound procedure
Mean difference in time taken to discharge patient from post-procedure recovery room | From end of endobronchial ultrasound procedure until final patient discharge from recovery room, assessed up to twelve hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Medicine, Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Kumari R, Jain K, Agarwal R, Dhooria S, Sehgal IS, Aggarwal AN. Fixed dexmedetomidine infusion versus fixed-dose midazolam bolus as primary sedative for maintaining intra-procedural sedation during endobronchial ultrasound-guided transbronchial needle aspiration: a double blind randomized controlled trial. Expert Rev Respir Med. 2021 Dec;15(12):1597-1604. doi: 10.1080/17476348.2021.1918000. Epub 2021 Apr 25. PMID 33849367